CLINICAL TRIAL: NCT04258449
Title: DOvEEgene Fleur: New Uterine Sampling Tool
Status: Recruiting | Type: Observational
Sponsor: McGill University (Other)
Collaborators: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other); GSE Biomedical (Other)
Responsible Party: Principal Investigator, Dr. Lucy Gilbert, Professor Department of Obstetrics & Gynecology and Department of Oncology, McGill University
Other Study IDs: 2020-6016
Record Dates: First submitted 2020-02-04; First posted 2020-02-06 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Women With Suspected or Confirmed Gynecological Disease
Keywords: Ovarian Cancer; Endometrial Cancer; Genomics; DNA tagging; Somatic mutations; Endometrial sampling; Uterine sampling; Medical device; Uterine biofluid
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Case: Participants must have suspected or confirmed upper genital tract cancer (uterine, tubal and ovarian) and must be scheduled to undergo surgery for tumor removal.
  Interventions: Device: DOvEEgene Fleur Sampling

INTERVENTIONS:
Device: DOvEEgene Fleur Sampling — Patients will undergo uterine sampling with DOvEEgene Fleur endometrial sampling device prior to surgical intervention, in addition to standard of care treatment.

SUMMARY:
This study is related to a previous study from the same group which started in 2014 (NTC02288676, McGill REB A08-M79-13B, MUHC REB 2020-5945) to develop a clinically implementable screening test -DovEEgene: developing and validating a novel molecular test for the early diagnosis of cancer of the endometrium, tubes and ovaries. This study is designed to identify endometrial, tubal and ovarian cancer very early based on identifying cancer-specific mutations (cancer DNA) in a pap sample taken from inside the uterus. The results are particularly encouraging given that control group is challenging with high background mutational burden from benign tumours, endometriosis, germ-line mutations etc.

To date, all the intrauterine samples were obtained using the commercially available TAO brush™ which is designed to take an endometrial sample. However, when patient tolerability was assessed using a numerical pain scale (NPS) ranging from 0 (no pain) to 10 (severe pain), patients rated the sampling using the TAO brush™ at 3.5 versus 0 for a cervical pap sample. These results were not surprising as the TAO brush™ was designed for dislodging strips of endometrial tissue to use for histopathologic examination. With respect to the investigators objective, which is to collect cancer cells that have exfoliated to the uterus, a sampler that collects these exfoliated cells with as little disturbance as possible to the underlying endometrium is preferred. In this sub-study, the investigators aim to evaluate a new endometrial sampling tool, the DOvEEgene Fleur, which is believe to be superior to the current TAO brush™ in terms of cancer detection, ease of use and patient tolerability. The sampler has been designed using materials/components found in the TAO brush™ and other approved medical devices.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age.
* Have capacity to understand the study.
* Be able to provide informed consent.
* If the patient has a recently treated cervical abnormality, she must have had a Pap smear with normal results at least 4 months following treatment by loop electrosurgical excision procedure (LEEP) or cone biopsy.
* Have suspected or confirmed cancer of the upper genital tract and be undergoing surgery for said tumor removal.

Exclusion Criteria:

* Prior hysterectomy.
* Be pregnant or possibly pregnant.
* Be nursing, as the device contains phthalates (plasticizers) that "have not been fully characterized and there may be concern for reproductive and developmental effects".
* Have an infected or inflamed cervix.
* Have a confirmed or suspected pelvic infection.
* Have a confirmed or suspected vaginal infection.
* Have had recent history of uterine perforation.
* Patients with recently treated cervical abnormalities must have a Pap smear with normal results at least 4 months following treatment by loop electrosurgical excision procedure (LEEP) or cone biopsy in order to be eligible.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participating hospital runs multiple weekly routine gynecologic oncology clinics. The cases include women scheduled to undergo surgery for tumor removal, for either proven or suspected upper genital tract cancer.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-12-11 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Patient related outcomes including pain and acceptability | up to 1 year
  Evaluate pain tolerability and acceptability during and after endometrial sample collection. This will be assessed using pain scores reported by participants on numeric pain scale (NPS) ranging from 0 to 10. Final pain scores with the DOvEEgene Fleur will be compared to historical pain scores collected with the TAO brush (Cook Medical).

SECONDARY OUTCOMES:
Feasibility of performing sample collection by clinicians | up to 1 year
  Ease of use of the DOvEEgene Fleur will be evaluated through a physician feedback form.
Quality/quantity of sample collection | up to 1 year
  Molecular assessment to verify DOvEEgene Fleur is capable of detecting cancer cells from the uterus.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Victoria Hospital (Glen Site), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gilbert L, Basso O, Sampalis J, Karp I, Martins C, Feng J, Piedimonte S, Quintal L, Ramanakumar AV, Takefman J, Grigorie MS, Artho G, Krishnamurthy S; DOvE Study Group. Assessment of symptomatic women for early diagnosis of ovarian cancer: results from the prospective DOvE pilot project. Lancet Oncol. 2012 Mar;13(3):285-91. doi: 10.1016/S1470-2045(11)70333-3. Epub 2012 Jan 17. PMID 22257524
- [Background] Kinde I, Bettegowda C, Wang Y, Wu J, Agrawal N, Shih IeM, Kurman R, Dao F, Levine DA, Giuntoli R, Roden R, Eshleman JR, Carvalho JP, Marie SK, Papadopoulos N, Kinzler KW, Vogelstein B, Diaz LA Jr. Evaluation of DNA from the Papanicolaou test to detect ovarian and endometrial cancers. Sci Transl Med. 2013 Jan 9;5(167):167ra4. doi: 10.1126/scitranslmed.3004952. PMID 23303603
- [Background] Gilbert L, Revil T, Meunier C, Jardon K, Zeng X, Martins C, Arseneau J, Fu L, North K, Schiavi A, Ehrensperger E, Artho G, Lee T, Morris D, Ragoussis J. The empress of subterfuge: cancer of the fallopian tube presenting with malapropism. Lancet. 2017 Sep 2;390(10098):1003-1004. doi: 10.1016/S0140-6736(17)31586-6. No abstract available. PMID 28872014
- [Background] Wang Y, Li L, Douville C, Cohen JD, Yen TT, Kinde I, Sundfelt K, Kjaer SK, Hruban RH, Shih IM, Wang TL, Kurman RJ, Springer S, Ptak J, Popoli M, Schaefer J, Silliman N, Dobbyn L, Tanner EJ, Angarita A, Lycke M, Jochumsen K, Afsari B, Danilova L, Levine DA, Jardon K, Zeng X, Arseneau J, Fu L, Diaz LA Jr, Karchin R, Tomasetti C, Kinzler KW, Vogelstein B, Fader AN, Gilbert L, Papadopoulos N. Evaluation of liquid from the Papanicolaou test and other liquid biopsies for the detection of endometrial and ovarian cancers. Sci Transl Med. 2018 Mar 21;10(433):eaap8793. doi: 10.1126/scitranslmed.aap8793. PMID 29563323
- See also: Parent study DOvEEgene: Diagnosing Ovarian and Endometrial Cancer Early Using Genomics (DOvEEgene) — https://clinicaltrials.gov/ct2/show/NCT02288676